CLINICAL TRIAL: NCT03973684
Title: Evaluation of Halitosis After Treatment With Photodynamic Therapy Randomized and Controlled Study
Brief Title: Evaluation of Halitosis After Treatment With Photodynamic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Phd, clinical professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: halitosis
Record Dates: First submitted 2019-05-21; First posted 2019-06-04 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2019-05

CONDITIONS: Halitosis
Keywords: bronchiectasis:; photodynamic therapy; periodontal disease; randomized controlled clinical study
MeSH Terms: conditions — Halitosis; Bronchiectasis; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: bio-equivalence study enrollment: 80
Who Masked: Participant, Investigator
Masking Description: Double (Participant ,investigator) Double Blind(Subject,Caregiver,Investigator,Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aPDT group (Active Comparator): G1- 40 patient 40 patients will be included in this group. One section of Pdt will be performed with the photosensitizer (PS). PS will be applied in sufficience quantity to cover the middle third and back of the tongue and wait for 5 minutes.six points with the distances of 1 cm between them will be irradiated. The apparatus shall be precalibrated at wavelength 660nm for 90 seconds per point.
  Interventions: Device: pdt experimental group; Other: tongue scraper group
- experimental tongue scrapper group (Experimental): 40 patients will be included in this group. Tongue scrapping will be performed by the same operator in all patients. Posterior -anterior movements will be performed with the scrapper over the lingual dorsum. in order to promote the mechanical removal of tongue coating
  Interventions: Device: pdt experimental group; Other: tongue scraper group

INTERVENTIONS:
Device: pdt experimental group — G1-40 patients Photodynamic therapy with methylene blue as photosensitizer
  device irradiation with low intensity laser (wave length = 660 nm) 9J (Jaules) per point(6 points) and radiant 90 seconds PS will be applied in sufficient quantity to cover the middle third and back of the tongue and wait for 5 minutes.six points with the distances of 1 cm between them will be irradiated.
Other: tongue scraper group — Tongue scrapping will be performed by the same operator in all patients. Posterior -anterior movements will be performed with the scrapper over the lingual dorsum. in order to promote the mechanical removal of tongue coating

SUMMARY:
Halitosis is the term used to define an unpleasant odor emanating from the mouth. Some lung diseases, such as bronchiectasis, are among the extra-oral causes of this condition. However, no studies have evaluated the reasons and treatment of halitosis in the population of adults with bronchiectasis. Methods and analysis: A randomized, controlled trial is proposed. Halitosis will be evaluated based on the measurement of volatile sulfur compounds (VSC) using gas chromatography. The participants (n=40) with halitosis and bronchiectasis will be randomized into two groups: G1-treatment with photodynamic therapy (n = 20) or G2-cleaning of the tongue with a tongue scraper (n = 20). After the treatments, a second evaluation will be performed, along with a microbiological analysis (qPCR) for the identification of the bacteria P. gingivalis and T. denticola. If the halitosis persists, the participants will receive periodontal treatment. The evaluation of halitosis and the microbiological analysis will be repeated. If the halitosis is solved, the participants will return after three months for an additional evaluation. This protocol will determine the effectiveness of phototherapy regarding the reduction of halitosis in healthy older adults and those with bronchiectasis.

DETAILED DESCRIPTION:
A single-center, randomized, controlled, single-blind clinical trial was designed in accordance with the criteria recommended for interventional trials in the SPIRIT Statement. The project for the proposed study received approval from the Human Research Ethics Committee o fNove de Julho University(certificate number: 1057901).

Selection of individuals - characterization of sample - Two groups will be composed of adults in treatment at the dental clinic of Nove de Julho University. After verbal and written explanations of the study, those who agree to participate will sign a statement of informed consent approved by the Human Research Ethics Committee of Nove de Julho University. The study will be conducted in compliance with the precepts stipulated in the Declaration of Helsinki (revised in Fortaleza, Brazil, 2013).

ELIGIBILITY:
Inclusion Criteria:

* every age in both genders
* With diagnosis of bronchiectasis (experimental group)
* Patients clinically stable (compensated) (control group)
* Have more than 10 teeth
* Do not have any changes in the anatomy of the back of the tongue (geographical or fissured tongue)
* With positive halitosis, SH2 level >112 ppb

Exclusion Criteria:

* Smokers or ex-smokers for less than 5 years
* Patients diagnosed with cystic fibrosis
* Patients with hypersensitivity to the photosensitizer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
halitmetry (gas chromatography test) | study completion an average of 1 year
  The portable Oral ChromaTM will be used for the assessment of halitosis. Oral air collection will follow the manufactured guide lines (Oral Chroma Manual Instruction). A syringe will be placed in the patient's mouth with the plunger completely inserted and the participant will breathe through the nose with the mouth closed for one minute.The plunger will then be withdrawn to fill the chamber with air. The gas injection needle will be placed on the syringe and the plunger will be adjusted to 0.5 ml. This air will be injected into the input of the device in a single motion. This procedure will be done before, immediately after aPDT or scraper and after periodontal treatment.

SECONDARY OUTCOMES:
microbiological analysis | before aPDT or scrapper , immediately after aPDT or scrapper , immediatly after periodontal treatment, 3 months later
  collecting biofilm sample from the region of the lingual dorsum with swab and identification of the bacteria P. gingivalis and T. denticola. Sample will be transferred to sterile tubes with tris-EDTA (Ethylenediamine tetraacetic acid). The analysis will be performed by PCR (polymerase Chain reaction) real time

OTHER OUTCOMES:
Oral Health Related Quality of life (OHRQoL) | before PDT or scrapper , 3 months after the halitosis treatment
  oral health related quality of life will be measured using halt (halitosis associated life quality test). The patient will respond 20 questions in a lickert point scale that ranges from 0 till 5, considering higher results as worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Carolina R Horliana, PhD, Principal Investigator — Nove de Julho University
Locations (1):
- Anna Carolina R.T. Horliana, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Schalch TO, Palmieri M, Longo PL, Braz-Silva PH, Tortamano IP, Michel-Crosato E, Mayer MPA, Jorge WA, Bussadori SK, Pavani C, Negreiros RM, Horliana ACRT. Evaluation of photodynamic therapy in pericoronitis: Protocol of randomized, controlled, double-blind study. Medicine (Baltimore). 2019 Apr;98(17):e15312. doi: 10.1097/MD.0000000000015312. PMID 31027098
- [Background] da Cunha Moraes G, Vitoretti LB, de Brito AA, Alves CE, de Oliveira NCR, Dos Santos Dias A, Matos YST, Oliveira-Junior MC, Oliveira LVF, da Palma RK, Candeo LC, Lino-Dos-Santos-Franco A, Horliana ACRT, Gimenes Junior JA, Aimbire F, Vieira RP, Ligeiro-de-Oliveira AP. Low-Level Laser Therapy Reduces Lung Inflammation in an Experimental Model of Chronic Obstructive Pulmonary Disease Involving P2X7 Receptor. Oxid Med Cell Longev. 2018 Mar 4;2018:6798238. doi: 10.1155/2018/6798238. eCollection 2018. PMID 29686745
- [Result] Costa-Santos L, Silva-Junior ZS, Sfalcin RA, Mota ACCD, Horliana ACRT, Motta LJ, Mesquita-Ferrari RA, Fernandes KPS, Prates RA, Silva DFT, Deana A, Bussadori SK. The effect of antimicrobial photodynamic therapy on infected dentin in primary teeth: A randomized controlled clinical trial protocol. Medicine (Baltimore). 2019 Apr;98(15):e15110. doi: 10.1097/MD.0000000000015110. PMID 30985667
- [Result] Isabella APJ, Silva JTC, da Silva T, Rodrigues MFSD, Horliana ACRT, Motta LJ, Bussadori SK, Pavani C, Silva DFTD. Effect of irradiation with intravascular laser on the hemodynamic variables of hypertensive patients: Study protocol for prospective blinded randomized clinical trial. Medicine (Baltimore). 2019 Apr;98(14):e15111. doi: 10.1097/MD.0000000000015111. PMID 30946378
- [Result] Ciarcia ACCDM, Goncalves MLL, Horliana ACRT, Suguimoto ESA, Araujo L, Laselva A, Mayer MPA, Motta LJ, Deana AM, Mesquita-Ferrari RA, Fernandes KPS, Bussadori SK. Action of antimicrobial photodynamic therapy with red leds in microorganisms related to halitose: Controlled and randomized clinical trial. Medicine (Baltimore). 2019 Jan;98(1):e13939. doi: 10.1097/MD.0000000000013939. PMID 30608426